CLINICAL TRIAL: NCT01407523
Title: An Open-label, Multicenter Study to Evaluate the Safety of Adjunctive Treatment With Intravenous Levetiracetam (L059 IV) in Epilepsy Patients Aged ≥ 16 Years With Partial Onset Seizures
Brief Title: An Open Label Study of L059 Intravenous (IV) in Japanese Epilepsy Subjects With Partial Onset Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01378
Record Dates: First submitted 2011-07-29; First posted 2011-08-02 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-01

CONDITIONS: Epilepsy; Partial Onset Seizures
Keywords: Levetiracetam; Infusion; Epilepsy; Partial Onset Seizures
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levetiracetam (Experimental): Twice daily intravenous (IV) infusion of Levetiracetam solution equivalent (mg-for-mg) to oral dose of Levetiracetam.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — * Formulation: concentrate for solution for infusion
  * Strength: Levetiracetam injection (100 mg/mL) will be packed in 5 mL glass vials (500 mg/5 mL)
  * Dosage: 1000 mg/day, 1500 mg/day, 2000 mg/day, 2500 mg/day or 3000 mg/day
  * Frequency: twice daily
  Other Names: Keppra®; E Keppra®

SUMMARY:
To evaluate the safety of Levetiracetam IV 15-minute infusion administered every 12 hours as adjunctive treatment in subjects with Partial Onset Seizures after switching from the equivalent Levetiracetam oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female aged ≥ 16 years
* Subject has Partial Onset Seizures that are classifiable according to the 1981 International League Against Epilepsy (ILAE) classification of Epileptic Seizures
* Subject weighs ≥ 40 kg
* Subject is currently taking Levetiracetam (LEV) as an adjunctive antiepileptic oral treatment with 1 to 3 other Antiepileptic Drugs (AEDs)

Exclusion Criteria:

* Subject has problems with venous accessibility
* Subject has participated in another clinical/pharmacological study during the last 4 weeks prior to the Screening Visit
* Subject is pregnant or lactating
* Subject has a history of suicide attempt(s) or presents with current depressive signs, current suicidal ideation, and/or behavior
* Subject has clinically significant Electrocardiogram (ECG) abnormalities according to the investigator

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (4):
- Japan (4):
  - 1, Niigata, Niigata
  - 2, Shizuoka, Shizuoka
  - 3, Kodaira, Tokyo
  - 4, Yamagata-city, Yamagata

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in July 2011 in order to end up with 4 centers in Japan.
  16 subjects were treated and completed the study. All 16 subjects are included in the Safety Set.
Pre-assignment Details: The Safety Set (SS) consisted of all subjects who started Levetiracetam intravenous (LEV IV) infusion after they had signed and dated the Informed Consent form. Participant Flow and Baseline Characteristics refer to the Safety Set (SS).
Groups:
- Levetiracetam: Twice daily intravenous (IV) infusion of Levetiracetam solution equivalent (mg-for-mg) to oral dose of Levetiracetam.
  Levetiracetam :
  * Formulation: concentrate for solution for infusion
  * Strength: Levetiracetam injection (100 mg/mL) will be packed in 5 mL glass vials (500 mg/5 mL)
  * Dosage: 1000 mg/day, 1500 mg/day, 2000 mg/day, 2500 mg/day or 3000 mg/day
  * Frequency: twice daily
Period: Overall Study
Arm/Group | Levetiracetam
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Levetiracetam
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Region of Enrollment [Number; unit: participants]
  Japan | 16
Weight [Mean (Standard Deviation); unit: kilogram] | 68.82 (12.38)
Height [Mean (Standard Deviation); unit: centimeter] | 163.40 (8.95)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events During the Entire Study Period (up to 32 Days)
Description: An Adverse Event (AE) is any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: During the entire Study Period from Screening (Day -14 to Day -1) over Evaluation Period (Day 1 to Day 4) to Follow-Up Period (Day 5 to Day 18)
Population: Safety Set (SS)
Measure: Number; unit: participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 16
participants | 5

2. Primary Outcome: Incidence of Treatment Emergent Serious Adverse Events During the Entire Study Period (up to 32 Days)
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that results in death, is life-threatening, results in significant or persistent disability/incapacity, is a congenital anomaly/birth defect (including that occurring in a fetus), or is an important medical event that may jeopardize the subject or may require medical or surgical intervention.
Time Frame: as for outcome 1
Population: Safety Set (SS)
Measure: Number; unit: participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 16
participants | 0

3. Secondary Outcome: Observed Plasma Trough Concentration of Levetiracetam Prior to Intravenous (iv) Infusion on Day 1
Description: Plasma sample for determination of Plasma trough concentration of Levetiracetam was taken prior to intravenous infusion of Levetiracetam in the morning of Day 1.
Time Frame: Day 1
Population: Pharmacokinetic Per Protocol Set (PK-PPS). This was defined as a subset of the Safety Set (SS) and consisted of subjects who had at least 1 evaluable Levetiracetam plasma concentration after intravenous administration. All 16 subjects from the SS are included in the PK-PPS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Levetiracetam
Number analyzed (Participants) | 16
micrograms per milliliter (µg/mL) | 11.732 (63.1)

4. Secondary Outcome: Observed Plasma Trough Concentration of Levetiracetam Prior to Intravenous (iv) Infusion on Day 4
Description: Plasma sample for determination of Plasma trough concentration of Levetiracetam was taken prior to intravenous infusion of Levetiracetam in the morning of Day 4.
Time Frame: Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Levetiracetam
Number analyzed (Participants) | 16
micrograms per milliliter (µg/mL) | 11.632 (59.6)

5. Secondary Outcome: Dose Normalized Plasma Trough Concentration of Levetiracetam Prior to Intravenous (iv) Infusion on Day 1
Description: Plasma sample for determination of Plasma trough concentration of Levetiracetam was taken prior to intravenous infusion of Levetiracetam in the morning of Day 1.
  Plasma trough concentration (Ctrough) was normalized to a dose of 500 mg as follows:
  Dose normalized Ctrough = Ctrough/last dose [mg] x 500 mg.
Time Frame: Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Levetiracetam
Number analyzed (Participants) | 16
micrograms per milliliter (µg/mL) | 6.611 (29.6)

6. Secondary Outcome: Dose Normalized Plasma Trough Concentration of Levetiracetam Prior to Intravenous (iv) Infusion on Day 4
Description: Plasma sample for determination of Plasma trough concentration of Levetiracetam was taken prior to intravenous infusion of Levetiracetam in the morning of Day 4.
  Plasma trough concentration (Ctrough) was normalized to a dose of 500 mg as follows:
  Dose normalized Ctrough = Ctrough/last dose [mg] x 500 mg.
Time Frame: Day 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Levetiracetam
Number analyzed (Participants) | 16
micrograms per milliliter (µg/mL) | 5.492 (29.4)

7. Secondary Outcome: Partial (Type 1) Seizure Frequency Per Day Over the Evaluation Period
Description: Partial (Type I) seizures can be classified into one of the following three groups: Simple partial seizures, Complex partial seizures, Partial seizures evolving to secondarily generalized seizures.
Time Frame: During the Evaluation Period (Day 1 to Day 4)
Population: Full Analysis Set (FAS). The FAS consisted of all subjects in the Safety Set (SS) with evaluable seizure frequency data over the Evaluation Period. All 16 subjects in the SS are included in the FAS.
Measure: Median (Inter-Quartile Range); unit: Seizures per day
Arm/Group | Levetiracetam
Number analyzed (Participants) | 16
Seizures per day | 0.38 [0.00 to 1.00]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over the entire Study Period from Screening (1 to 14 days prior to the first intravenous infusion) over Evaluation Period (4 days) to the end of Follow-Up Period (1 to 14 days after the final intravenous infusion).
Description: AEs refer to Safety Set (SS). The Safety Set (SS) consisted of all subjects who started Levetiracetam intravenous (LEV IV) infusion after they had signed and dated the Informed Consent form.
Arm/Group | Levetiracetam
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 5/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=16)
Gingivitis (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Injection site inflammation (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Injection site swelling (General disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days